CLINICAL TRIAL: NCT00028405
Title: A Multicenter Phase I Safety and Tolerability Study of the Oncolux System for Intratumoral Delivery of Non-Coherent Light for the Photoactivation of LS 11 in Patients With Refractory Solid Tumors
Brief Title: Photodynamic Therapy System for Patients With Refractory/Unresponsive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Light Sciences LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSC-OL001; NCT00049205 (obsolete NCT alias)
Record Dates: First submitted 2002-01-04; First posted 2002-01-09 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: Liver Metastasis; Pelvic Cancer; Head and Neck Cancer; Sarcoma; Rectal Cancer; Breast Cancer; Colorectal Cancer; Mouth Cancer
Keywords: Photodynamic Therapy; Bulky Tumor; Refractory Tumor; Head and Neck Cancer; Breast Cancer; Pelvic Tumors; Liver Metastasis; Colorectal Cancer; Sarcoma; Anal Cancer; Oral Cancer; Recurrent; Lymphadenopathy; Ovarian Cancer; Cervical Cancer
MeSH Terms: conditions — Pelvic Neoplasms; Head and Neck Neoplasms; Sarcoma; Rectal Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Mouth Neoplasms; Neoplasms; Anus Neoplasms; Recurrence; Lymphadenopathy; Ovarian Neoplasms; Uterine Cervical Neoplasms

INTERVENTIONS:
Drug: LS 11(Taporfin Sodium)
Device: Lumaflex Light Delivery Catheter

SUMMARY:
This multi-center photodynamic therapy study plans to treat patients with large tumors in any superficial location, sarcoma, tumors of oral/oro-pharyngeal cavity, tumors with extensive pelvic involvement, or liver metastasis. The treatment is limited to patients that have failed to respond to currently approved methods of treatment. The study involves a single, intravenous administration of an investigational drug, LS11 (previously studied in approximately 80 cancer patients) and the placement of a novel, flexible light delivery catheter inside the tumor by a minor surgical procedure. The activation of LS11 by the light delivery catheter over a period of 1-24 hrs may result in destruction of tumor tissue.

DETAILED DESCRIPTION:
In this Phase I photodynamic therapy study, patients will undergo a standard CT scan to determine the suitability of the treatment. In those patients that qualify the entry criteria, a light delivery catheter will be directly inserted in the tumor through a minor surgical procedure. The patients will then be injected with the photosensitive drug, LS11. One hour following the drug injection, light energy will be delivered from the light delivery catheter for a period of 1-24 hours. The duration of the light treatment for a given patient may be based on various factors including when a given patient enters the study. Following the delivery of light energy, the light delivery catheter will be removed from the tumor. The insertion and removal of the catheter will be carried out under the guidance of CT scan. The patients will be asked to take precautions from external light exposure for a period of time. The patients will undergo CT scan and other tests on days 7, 14 and 42 to evaluate safety of the treatment, tumor cell death and treatment response. Blood samples will be taken at different time points to examine the clearance of the drug from the body.

ELIGIBILITY:
Primary Inclusion Criteria:

* Target tumors accessible for percutaneous implantation under CT (and ultrasound if needed) guidance in any superficial location, sarcoma, tumors of oral/oro-pharyngeal cavity, tumors with extensive pelvic involvement, or liver metastasis.
* Patient has failed prior surgery or chemotherapy or radiation therapy and the tumor is refractory.
* Tumor mass is not immediately adjacent to, or directly invading a major vessel or hollow viscus such that tumor necrosis could result in hemorrhage or perforation.
* Patient has not received prior chemotherapy for at least 4 weeks and patient has recovered from toxicity.
* Patient has an ECOG performance status of 0-3 (Karnofsky 30 or higher).
* If patients have received radiotherapy to sites of disease other than the one planned for insertion of the light delivery catheter, then the patient must have no current local or systemic toxicity from the prior radiation.
* Patient has recovered from all previous surgery in the judgment of the Principal Investigator.
* Patient has not been treated with any biologics (excluding hormones) at least 4 weeks prior to the screening and patient has recovered from any toxicity.
* Age 18 or older.
* Minimum life expectancy of 12 weeks.
* Ability to provide informed consent.
* All tumors must:

  * have a minimum dimension that exceeds 4 x 2.8 cm;
  * have a shape and location such that the mid-point on the light delivery catheter will be greater than 2.0 cm from any structure which, if damaged by PDT treatment, would result in pain or injury to the patient.

Exclusion Criteria:

* History of cardiovascular abnormalities, including, myocardial infarction in the last 6 months, arrhythmias, uncontrolled congestive heart failure;
* History of ongoing, significant active medical illness that might create a risk for the patient, in the opinion of the Investigator;
* History of known or suspected porphyria;
* Concomitant use of other drugs known to produce skin photosensitivity;
* Women who are pregnant or lactating;
* Hematopoietic abnormalities from the baseline examination, as evidenced by the following laboratory values (US Units):Hemoglobin <10 g/dL; White blood cell (WBC) count <2500/mm3;Neutrophil count < or = 1500/uL;Platelet count < or = 100,000/mm3;
* Renal or liver function abnormalities from the baseline examination, as evidenced by the following laboratory values(US Units):Serum Creatinine >2.0 mg/dL;Total bilirubin > 2.0 mg/dL; SGOT (AST) > 3x the ULN;SGPT (ALT) > 3x the ULN; GGT> 3x the ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2001-11; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Jay Winship, MD, Study Director — Sr. Vice President of R & D and Chief Medical Officer
Locations (6):
- United States (6):
  - University of Arizona, VA Medical Center, Tucson, Arizona
  - Detroit Medical Center, Wayne State University, Detroit, Michigan
  - East Carolina State University, Brody School of Medicine, Greenville, North Carolina
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Background] Taber SW, Fingar VH, Coots CT, Wieman TJ. Photodynamic therapy using mono-L-aspartyl chlorin e6 (Npe6) for the treatment of cutaneous disease: a Phase I clinical study. Clin Cancer Res. 1998 Nov;4(11):2741-6. PMID 9829737
- See also: Related Info — http://www.Lightsciences.com